CLINICAL TRIAL: NCT02492308
Title: Effect of Autologous Stromal Vascular Fraction Derived Mesenchymal Stem Cell in Living-Related Kidney Transplants: A Randomized Controlled Trial
Brief Title: Induction With SVF Derived MSC in Living-related Kidney Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVF-LR
Record Dates: First submitted 2015-07-04; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Living-relative Kidney Transplantation
Keywords: kidney; transplantation; MSC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SVF-MSC induction (Experimental): 1. collection of autologous SVF
  2. culture of SVF to abstain MSC
  3. infusion of MSC during and after living-relative kidney transplantation
  Interventions: Procedure: SVF-MSC induction
- Basiliximab induction (Active Comparator): The control group will be inducted with Basiliximab
  Interventions: Drug: Basiliximab induction

INTERVENTIONS:
Procedure: SVF-MSC induction — Procedure: infusion of autologous SVF derived MSC to the recipients of living-relative kidney transplant.
  Subjects with uremia in the intervention group will undergo puncture to collect SVF, then SVF will be cultured to abstain MSC, and the abstained MSC will be infused to the recipients during kidney transplant operation and on 7, 14, and 21 POD
  Arms: SVF-MSC induction
Drug: Basiliximab induction — The control group will be inducted with Basiliximab before living-relative kidney transplantation and on POD 4
  Arms: Basiliximab induction

SUMMARY:
The objective of this trial is to determine if autologous SVF derived MSC can effectively reduce the need for post transplant immunosuppressant in living-relative kidney transplantation. 120 patients eligible for the study as described below will be enrolled, with 60 patients in intervention group and 60 in control group.

DETAILED DESCRIPTION:
The objective of this trial is to determine if autologous SVF derived MSC can effectively reduce the need for post transplant immunosuppressant in living-relative kidney transplantation. Emphasis will be placed on the safety of autologous SVF derived MSC infusion, dosage of immunosuppressant, GFR, percentage of acute rejection. 120 patients eligible for the study as described below will be enrolled, with 60 patients in intervention group and 60 in control group. In interventional group we will collect SVF from recipients with special instruments before transplantation, and culture SVF to abstain MSC. The abstained MSC will be infused to the recipients of living-relative kidney transplantation during operation and on 7, 14, 21 POD. We will assess whether induction therapy with autologous SVF derived MSC is feasible in living-relative donor kidney transplantation. The effectiveness of autologous SVF derived MSC induction therapy on reducing of immunosuppressant, reducing the rate of rejection, elevating patient and allograft survival, improving allograft function from day 0 to 12 months after transplantation. Additionally, we will assess the percentage of acute rejection or antibody mediated rejection by Banff criteria, the incidence of delayed graft function (defined as the need for post-transplant dialysis within one week), and the incidence of adverse events including infection, grade 3 and above non-hematologic toxicities, and grade 4 hematologic toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Uremia patient of any race that is greater than or equal to 18 years of age but less than 60 years old 2. Patient is willing to receive a kidney from a certifiable living-relative donor 18-60 years of age 3. Patient is willing and capable of giving written informed consent for study participation and able to participate in the study for 12 months

-

Exclusion Criteria:

1. Women who are pregnant, intend to become pregnant in the next 1 years, breastfeeding, or have a positive pregnancy test on enrollment or prior to study medication administration
2. Patient with prior solid organ transplant or cell transplant (e.g. bone marrow or islet cell).
3. Patient is deemed likely to have a second solid organ transplant or cell transplant (e.g. bone marrow or islet cell) in next 3 years
4. Patient receiving a concurrent SOT (heart, liver, pancreas)
5. ABO incompatible donor recipient pair or CDC crossmatch positive transplant
6. Sensitized patients (most recent anti-HLA Class I or II Panel Reactive Antibodies (PRA)>10% by a CDC-assay) or patients identified a high immunological risk by the transplant physician
7. Donors with cardiac death (non-heart beating donor) 8 Donors or recipients are known hepatitis C antibody-positive or polymerase chain reaction (PCR) positive for hepatitis C

9. Donors or recipients are known hepatitis B surface antigen-positive or PCR positive for hepatitis B 10. Donors or recipients are known human immunodeficiency virus (HIV) infection 11. Recipients at risk for tuberculosis (TB)

1. Current clinical, radiographic or laboratory evidence of active or latent TB as determined by local standard of care
2. History of active TB:

(I). Within the last 2 years, even if treated (II) Greater than 2 years ago, unless there is documentation of adequate treatment according to locally accepted clinical practice c. Recipients at risk of reactivation of TB precludes administration of conventional immunosuppressant (as determined by investigator and based upon appropriate evaluation) 12. Recipients with any significant infection or other contraindication that would preclude transplant 13. Recipients with a history of hypercoagulabale state 14. Recipients with a history of substance abuse (drugs or alcohol) within the past 6 months, or psychotic disorders that are not capable with adequate study follow-up.

15. Recipients with active peptic ulcer disease (PUD), chronic diarrhea, or gastrointestinal problem affect absorption 16. Recipients with a history of cancer within the last 5 years (exception: non-melanoma skin cell cancers cured by local resection are permitted) 17. Recipients with a chest radiograph (no more than 2 months prior to randomization) consistent with an acute lung parenchymal process and malignancy 18. Recipients with a hypersensitivity to any study drugs 19. Recipients who have used any investigational drug within 30 days prior to the Day 1 visit 20. Prisoner or patients compulsorily detained (involuntarily incarcerated) for treatment or either a psychiatric or physical (e.g. infectious disease) illness

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Effects of autologous SVF derived MSC transplantation on reducing the dosage of immunosuppressant in living-related kidney transplant recipients. | 1 year
  Reducing the dosage of immunosuppressant by 30% of CNI in living-related kidney transplant recipients.

SECONDARY OUTCOMES:
Changes in renal function | 1 year
  • Changes in renal function as determined by estimated glomerular filtration rate (eGFR) and proteinuria (>1g) at 1 year post transplant
Incidence of acute rejection | 1 year
  Incidence of acute rejection (biopsy confirmed acute rejection according to Banff creteria)
Incidence of delayed graft function | 1 month
  Incidence of delayed graft function (defined as need for post-transplant dialysis within one week)
Allograft survival | 1 year
  Allograft survival at 1 year post transplant
Infection adverse event | 1 year
  Incidence of death, allograft loss, and hospitalization due to infection at 1 year.
Non-hematologic toxicities | 1 year
  Incidence of grade 3 and above non-hematologic toxicities
Hematologic toxicities | 1 year
  Incidence of grade 4 hematologic toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Tan Jianming, MD PhD, Study Director — Fuzhou General Hospital, Xiamen Univ
Locations (1):
- Xi er huan road No.156, Fuzhou, Fujian, China